CLINICAL TRIAL: NCT04141813
Title: The Effects of the Pilgrimage in the Way of Saint James on Mental Health and Well-being (ULTREYA Project)
Brief Title: The Effects of the Pilgrimage in the Way of Saint James on Mental Health and Well-being (ULTREYA)
Acronym: ULTREYA
Status: Completed | Type: Observational
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Universidad de Zaragoza (Other); Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Juan Vicente Luciano, Principal Investigator, Fundació Sant Joan de Déu
Other Study IDs: PIC-141-19
Record Dates: First submitted 2019-10-22; First posted 2019-10-28 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Pilgrimage
Keywords: mindfulness; mental health; well-being; peregrination; walking; forest-bathing; outdoor therapy; wilderness therapy; adventure therapy
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pilgrims doing the "Camino de Santiago" (any route): In the present study we utilized the "Ultreya" dataset. The Ultreya study is an online longitudinal study aimed at evaluating the effects of the pilgrimage on the Way of Saint James on mental health and wellbeing (www.estudiocamino.org). This pilgrimage involves hundreds of paths around Europe with a common termination at Santiago de Compostela (Spain), and it was one of the most important Christian pilgrimages during the Middle Ages. Currently, it is walked by thousands of people (>300,000 per year).

SUMMARY:
Objectives: This study aims to evaluate the effects of pilgrimage to Santiago de Compostela on mood, satisfaction with life, happiness, ability to pay attention to the present moment and the capacity to make choices in a more conscious and values-oriented way. Other personal aspects that could be related to the effects of the Camino and that may also mediate some of its effects (e.g., personal reasons for walking, socialization along the Camino, number of days walked, physical pain associated with walking, previous pilgrimages to Santiago, etc.) will be also assessed.

Methods: This is a naturalistic study with a 3-month follow-up. Voluntary participation of pilgrims doing one of the "Way of Saint James" routes will be requested. Participants will be asked to complete an online questionnaire with sociodemographic data and outcome measures (e.g. mindfulness, satisfaction with life, depression, stress, anxiety) before starting the Camino, at the end of the Camino and 3 months later. These evaluations will help us discover the effects of the Camino de Santiago on mental health and well-being in the short- and mid-term.

For more information (and/or to participate), go to: http://estudiocamino.org/

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years old)
* Willing to go on pilgrimage in the Way of Saint James
* With or without previous experience in this pilgrimage
* Walking or cycling in the pilgrimage
* Finishing or not at "Santiago de Compostela"
* Ability to understand and read Spanish or English
* With internet access (via PC or smatphone)
* With signed informed consent to participate in the present study

Exclusion Criteria:

* Not walking for 4 or more days
* With incomplete baseline data
* With baseline/post assessments >1 month previous starting/ending the pilgrimage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pilgrims in the Way of Saint James.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire, short form (PHQ-2; Kroenke, Spitzer, & Williams, 2003) | Through study completion, an average of 3 months
  PHQ-2 is a 2-item measure assessing frequency of the two core depression symptoms (depressed mood and anhedonia) over the past two weeks, using a 4-point Likert scale (from 0= "not at all" to 3= "nearly every day"; total score ranges from 0 to 6). Higher scores indicate greater depressive symptoms.
General Anxiety Disorder scale, short form (GAD-2, Kroenke, Spitzer, Williams, Monahan, & Löwe, 2007) | Through study completion, an average of 3 months
  GAD-2 is a 2-item scale that serves as an initial screening tool for generalized anxiety. Items are on a 4-point Likert scale (from 0= "not at all" to 3= "nearly every day"; total score ranges from 0 to 6). Higher scores indicate greater anxiety symptoms.
Perceived Stress Scale, short form (PSS-4; Cohen, Kamarck, & Mermelstein, 1983) | Through study completion, an average of 3 months
  PSS-4 is a 4-item scale which measures the degree to which respondents appraised situations as stressful in the last month. Responses are scored on a Likert-scale between 0 = "never" and 4 = "very often" (total score ranges from 0 to 16). Higher scores indicate greater perceived stress.
Satisfaction with Life Scale (SWLS; Diener, Emmons, Larsen, & Griffin, 1985) | Through study completion, an average of 3 months
  SWLS assesses global life satisfaction. It contains five items rated on a 7-point Likert scale ranging from 1 ("strongly disagree") to 7 ("strongly agree") ( total scores range from 5 to 35). Higher scores indicate greater perceived satisfaction with life/wellbeing.
Subjective Happiness Scale (SHS; Lyubomirsky & Lepper, 1999) | Through study completion, an average of 3 months
  SHS is a measure of global subjective happiness and consists of four items with a 7-point Likert-type scale. Mean total score ranges from 1 to 7, with greater scores indicating higher levels of perceived happiness.
International Positive and Negative Affect Schedule, short form (I.PANAS-SF; Thompson, 2007) | Through study completion, an average of 3 months
  I-PANAS-SF is a 10-item version of the International Positive and Negative Affect Schedule (PANAS) to measure positive and negative affect. Items are on a 5-point scale that ranges from "never" (1) to "always" (5). Subscale scores (i.e. Positive affect or Negative affect) may range from 5 to 25 with higher scores meaning greater presence of positive or negative affect .

SECONDARY OUTCOMES:
Five Facet Mindfulness Questionnaire, 15-item form (FFMQ-15; Baer et al., 2012) | Through study completion, an average of 3 months
  FFMQ-15 measures trait-like tendency to be mindful in daily life and comprises five different facets with three items each (i.e. Observe, Describe, Act with Awareness, Nonreact, Nonjudge). Items are answered on a 5-point Likert-scale ranging from 1 ("never or very rarely true") to 5 ("very often or always true") with subscale scores ranging from 3 to 15. Higher scores indicate greater dispositional mindfulness.
Nonattachment Scale, short form (NAS-7; Elphinstone, Sahdra, & Ciarrochi, 2014) | Through study completion, an average of 3 months
  The NAS-7 is a 7-item measure scored on a 6-point scale ranging from 1 = disagree strongly to 6 = agree strongly and designed to measure nonattachment. Its scores range from 7 to 42, with higher scores indicating greater nonattachment.
Engaged Living Scale (ELS; Trompetter et al., 2013) | Through study completion, an average of 3 months
  The ELS is a 16-item scale, with each item rated on a five-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree). It comprises two subscales: Valued Living (10 items; scores ranging from 10 to 50) and Life Fulfillment (6 items; with scores ranging from 6 to 30). Higher scores indicate greater perceived valued living or life fulfillment.

CONTACTS AND LOCATIONS:
Overall Officials: Javier García-Campayo, PhD, Principal Investigator — Universidad de Zaragoza; Joaquim Soler, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Marcelo Demarzo, PhD, Principal Investigator — Univesidad Federal de Sao Paulo; Manu Mariño, MSc, Principal Investigator — Quietud Mindfulness Centre; Jesús Montero-Marin, PhD, Principal Investigator — Dharamsala Institute of Mindfulness and Psychotherapy; Albert Feliu-Soler, PhD, Principal Investigator — Fundació Sant Joan de Déu; Juan V Luciano, PhD, Principal Investigator — Fundació Sant Joan de Déu
Locations (1):
- Teaching, Research & Innovation Unit - Parc Sanitari Sant Joan de Déu, Sant Boi de Llobregat, Barcelona, Spain

REFERENCES:
- See also: Study website — http://www.estudiocamino.org/
- See also: Ultreya project (Researchgate) — https://www.researchgate.net/project/ULTREYA-PROJECT-The-effects-of-the-pilgrimage-to-Santiago-Way-of-Saint-James-on-mindfulness-mental-health-and-well-being